CLINICAL TRIAL: NCT04954248
Title: Pilot Study for Simultaneous PET-MR Imaging of Covid-19 Associated Neurological Complications Using a Brain Dedicated PET Insert
Brief Title: Pilot Study for PET/MR Imaging of Covid-19
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The associated funding source was ended, and the proposed duration of the study ended.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Craig Levin, Professor, Radiology/Nuclear Medicine, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-59616
Record Dates: First submitted 2021-07-07; First posted 2021-07-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Brain Diseases; Covid19
MeSH Terms: conditions — Brain Diseases; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Covid-19 Negative/Uninfected Population (Experimental): 5 participants will be recruited, injected with radiopharmaceutical, and imaged on the 3T PETMR with PET insert.
  Interventions: Diagnostic Test: Injected radiotracer with PET Insert
- Covid-19 Positive/Infected Population (Experimental): 5 participants will be recruited, injected with radiopharmaceutical, and imaged on the 3T PETMR with PET insert.
  Interventions: Diagnostic Test: Injected radiotracer with PET Insert

INTERVENTIONS:
Diagnostic Test: Injected radiotracer with PET Insert — 1. Informed consent will be obtained before beginning any study procedures.
  2. Participants will receive a small quantity of an FDA approved radiotracer. The PET insert is placed within a 3T MRI scanner, where PET and MRI imaging will be completed.

SUMMARY:
The primary goal of this project is to study the feasibility of a prototype brain-dedicated PET insert for an MR scanner for simultaneous acquisition of PET/MR images of metabolism and perfusion in Covid-19 negative and positive/once positive subjects. This study serves as a pilot study for establishing an imaging protocol for combined PET and MR derived functional information as well as MRI acquired anatomical information.

DETAILED DESCRIPTION:
This study is a non-randomized non-treatment study. The intention of this work is an assessment of the PET insert technology, and not, for example, to perform a treatment assessment or drug assessment. This work will actively recruit 10 individuals (5 Covid-19 negative and 5 Covid-19 previously positive in the last 180 days) to perform imaging of the brain with an FDA-approved radiotracer.

ELIGIBILITY:
Inclusion Criteria:

1. Whole body radiation dose in the last year of less than 5000 mrem determined via subject verbal history reporting
2. Must be at least 21 years of age
3. Deemed healthy to endure duration of imaging study as confirmed via study PI
4. Proof of COVID-19 viral or antibody testing within the timeframe of >20 days but <=180 days prior to scan.

Exclusion Criteria:

1. History of non-MRI compatible surgeries, implants, or activities
2. Pregnant or nursing
3. History of allergic reactions to PET radiotracers (via patient verbal report and /or medical record review.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-08-19 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
PET/MR | Up to 24 months
  The key specific measurement is the resulting PET/MR image obtained from the single subject scan.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Levin, M. Phil., PhD., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States